CLINICAL TRIAL: NCT00211276
Title: A Phase II Multicenter Study of ONTAK in Patients With Relapsed or Refractory, B-Cell Non-Hodgkins Lymphoma.
Brief Title: A Study of ONTAK in Patients With Relapsed or Refractory, B-Cell Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #123
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — denileukin diftitox

INTERVENTIONS:
Drug: ONTAK (denileukin diftitox)

SUMMARY:
The goal of this clinical research study is to find out if the study drug, ONTAK (denileukin diftitox), can shrink or slow the growth of B-cell non-Hodgkin's lymphoma (NHL) in patients whose disease has not responded to prior treatments, or has relapsed after an initial response to prior treatments. The safety of treatment with ONTAK will also be studied. The hypothesis is that patients with relapsed or refractory B-cell NHL and mild to moderate myelosuppression treated with ONTAK at a new dosing regimen will respond sufficiently to warrant further study.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory B-Cell NHL
* Histological documentation of diffuse large B-cell lymphoma, follicular lymphoma (grade 1, 2, or 3), small lymphocytic lymphoma or transformed B-Cell lymphoma.
* Bi-dimensionally measurable disease with at least one lymph node or tumor mass measuring > or equal to 4 cm2
* ECOG performance status less than or equal to 2.
* Failure to respond or progression of disease after 2 or more prior treatment regimens; this may include high dose therapy (HDT) with stem cell transplantation (SCT). Patients with prior HDT plus SCT will be considered as having "diminished bone marrow reserve"
* At least 18 years of age
* At least 3 weeks from last anti-lymphoma therapy
* Mild to moderate cytopenia defined as any of the following:
* ANC > or equal to 1,000/microL and < 1,500/microL off growth factors
* WBC counts > or equal to 2,000/microL and < 4,000/microL off growth factors or
* Platelet count > or equal to 40,000/microL (25,000/microL if thrombocytopenia is secondary to marrow involvement by lymphoma) and < 150,000/microL.
* Acceptable organ function defined as all of the following:
* Bilirubin < or equal to 1.5 times the upper limit of normal (ULN)
* SGOT (AST) and SGPT (ALT) < or equal to 2 times the ULN.
* Serum creatinine < 2 times ULN.
* Serum albumin > or equal to 3.0 g/dL
* Female patient of childbearing potential must have a negative pregnancy test within seven days prior to study drug administration, and must agree to use an effective means of contraception throughout the study.
* Life expectancy of at least 16 weeks.
* Patients must have reviewed, signed and dated a witnessed informed consent document that has been approved by the IRB of each participating center.

Exclusion Criteria:

* Less than 6 months from prior allogeneic stem cell transplant and/or patient with active graft versus host disease (GVHD) Grade > or equal to 2.
* Prior history of veno-occlusive disease of the liver.
* Inability to comply with protocol requirements of this study for intravenous administration of ONTAK.
* Pregnant women or lactating women who are breastfeeding or women planning to become pregnant during the treatment period.
* Serious intercurrent medical illnesses or active infections that, in the investigators opinion, might interfere with the interpretation of the study safety data or compromise the patients ability to carry out the treatment program.
* Known history of seropositivity for HIV or chronic hepatitis (testing for HIV is not required).
* Known hypersensitivity to ONTAK or any of its components: diptheria toxin, interleukin-2 or excipients.
* Experimental therapy within 4 weeks prior to study entry.
* Patients diagnosed with congestive heart failure, NYHA Class III or IV, ventricular tachycardia, fibrillation, or a history of myocardial infarction in the 12 months prior to study entry.
* Any prior radiation therapy within four weeks of enrollment, or prior radiation therapy to the only site of evaluable disease unless disease progression has occurred in that site.
* Patients on concurrent corticosteroids as treatment for NHL. The use of tapering doses or low doses of corticosteroids for resolving GVHD, or the use of corticosteroids as premedication prior to ONTAK or as a transient treatment for hypersensitivity reactions is permitted as necessary.
* History of prior malignancy within the preceding 5 years, except for successfully treated cervical carcinoma in situ or basal cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Disease Response will be evaluated by CT or MRI scans at baseline, every 8 weeks while on therapy, and every 3 months after therapy, using standard response criteria defined by Cheson et al.

SECONDARY OUTCOMES:
Safety data will include laboratory, history and physical, and adverse events reports for both local and systemic signs or symptoms of study patients. Survival at one year post-therapy will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Myron Czuczman, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (12):
- United States (12):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Pacific Coast Hematology/Oncology, Fountain Valley, California
  - University of California, Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania